CLINICAL TRIAL: NCT06114498
Title: Hospital Register of Decompensated Heart Failure With Preserved Ejection Fraction
Status: Active, not recruiting | Type: Observational
Sponsor: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Collaborators: Moscow State Clinical Hospital named after V.V. Veresaev (Unknown)
Responsible Party: Sponsor
Other Study IDs: 04-05/23
Record Dates: First submitted 2023-10-28; First posted 2023-11-02 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Obesity, Mild; Decompensated Heart Failure
Keywords: Hearth failure; Decompensated Heart Failure; Heart Failure with Preserved Ejection Fraction; HFpEF; Heat shock protein; Obesity
MeSH Terms: conditions — Obesity; Lymphoma, Follicular | interventions — Echocardiography; Fluorescence Polarization Immunoassay

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient with HFpEF with decompensation: 120 patients hospitalized with a clinical picture of acute decompensation of heart failure (shortness of breath, orthopnea, clinical signs of "cardiac asthma" and/or "pulmonary edema") in the city clinical hospital named after. V.V. Veresaeva, Moscow. Patients with a confirmed diagnosis in accordance with instrumental and/or laboratory criteria
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: Bioimpedance; Diagnostic Test: Immunoassay; Diagnostic Test: Routine biochemistry
- Control group: 40 particularly healthy people without heart failure and acute cardiovascular diseases
  Interventions: Diagnostic Test: Bioimpedance; Diagnostic Test: Immunoassay; Diagnostic Test: Routine biochemistry

INTERVENTIONS:
Diagnostic Test: Echocardiography — Transthoracic echocardiography at rest: with determination of epicardial fat tissue thickness, intensity of mitral regurgitation.
  Groups: Patient with HFpEF with decompensation
Diagnostic Test: Bioimpedance — Bioelectrical impedance analysis research
Diagnostic Test: Immunoassay — Enzyme immunoassay of heat shock proteins in blood serum
  Other Names: ELISA
Diagnostic Test: Routine biochemistry — Measuring of routine biochemical parameters (glucose, total protein, creatinine, urea, uric acid, total bilirubin, direct bilirubin, total cholesterol, triglycerides, low and high density lipoprotein cholesterol, Lactate dehydrogenase, creatine phosphokinase, aspartate aminotransferase, alanine aminotransferase, sodium, potassium and special (C-reactive protein, N-terminal pro b-type natriuretic peptide)

SUMMARY:
Study Aim is creation of the Hospital Register of patients with heart failure with preserved ejection fraction (HFpEF) for a comprehensive assessment of the influence of gender characteristics, clinical and anamnestic factors, body composition, topical characteristics of congestion, instrumental data and markers of cellular inflammation and stress on immediate and long-term outcomes in patients with acute decompensated heart failure with preserved ejection fraction.

During the study it is planned to assess gender, clinical and anamnestic indicators preceding hospitalization of patients in the hospital; characterize the features of comorbid status in the studied group of patient; study the features of drug therapy at the prehospital stage and during hospitalization in the study group of patient; assess adverse hospital outcomes and outcomes 6 months after hospital discharge and identify factors associated with them; assess body composition in patients with acute decompensated heart failure with preserved ejection fraction in obese patients upon admission to the hospital; characterize the severity and topical characteristics of congestion and compare with the phenotypes of acute decompensation of heart failure; asess adverse in-hospital outcomes and outcomes 6 months after hospital discharge and identify factors associated with them; conduct a clinical and instrumental examination of patients diagnosed with compensated and decompensated HFpEF, verified by echocardiography at rest, as well as in patients with HFpEF verified after an additional diastolic stress test with assessment of intracardiac hemodynamic; analyze the serum concentrations of biochemical markers associated with cellular stress in these groups of patients, as well as in the control group of apparently healthy people; conduct an analysis of associations of biomarker levels with clinical characteristics of patients, the presence of comorbid diseases, including obesity, as well as with data from instrumental examination methods; assess the diagnostic capabilities of HFpEF, defined by various criteria, based on the concentration of the new biomarkers The results obtained will allow us to evaluate the characteristics of the course and outcomes of the disease in Moscow patients, depending on the phenotype of acute decompensation of HFpEF, hospitalized in the hospital during the study period. It is expected to identify phenotypes of acute decompensation of HFpEF that affect the duration of hospitalization and the development of adverse outcomes in the hospital and long-term period of the disease.

DETAILED DESCRIPTION:
THE RELEVANCE OF RESEARCH Identifying patients with heart failure with preserved ejection fraction (HFpEF) represents a significant public health challenge. In a significant proportion of patients with HFpEF, no specific underlying etiology has been identified, with the exception of cardiovascular risk factors such as hypertension, obesity, diabetes mellitus, the presence of atrial fibrillation, and others. Many of these patients are classified as having hypertension and do not receive the necessary amount of preventive interventions aimed at reducing hospitalizations and increasing life expectancy. The incidence of hospitalization for acute decompensated heart failure is increasing, mainly due to acute HFpEF. It is hypothesized that systemic inflammation resulting from comorbidities such as obesity, diabetes mellitus, and hypertension is responsible for the pathogenesis of myocardial structural and functional changes in HFpEF. Therefore, assessment of clinical and anamnestic factors and their relationship with signs of structural changes, functional disorders of intracardiac hemodynamics, signs of congestion and systemic inflammation will help optimize the diagnostic and treatment algorithm for patients with acute decompensation of HFpEF.

In this context, additional markers such as body composition measures, ultrasound congestion criteria, and cellular stress-related biomarkers may complement or even surpass traditional markers in predicting the severity and prognosis of HFpEF.

The creation of a register and analysis of the data entered into it will help improve the comprehensive diagnosis of decompensated HFpEF

PURPOSE OF THE STUDY:

Creation of a register of patients with HFpEF for a comprehensive assessment of the influence of gender characteristics, clinical and anamnestic factors, body composition, topical characteristics of congestion, instrumental data and markers of cellular inflammation and stress on immediate and long-term outcomes in patients with acute decompensated heart failure with preserved ejection fraction.

During the study it is planned

1. Assess gender, clinical and anamnestic indicators preceding hospitalization of patients in the hospital.
2. Characterize the features of comorbid status in the studied group of patients.
3. To study the features of drug therapy at the prehospital stage and during hospitalization in the study group of patients.
4. Assess adverse hospital outcomes and outcomes 6 months after hospital discharge and identify factors associated with them.
5. To assess body composition in patients with acute decompensated heart failure with preserved ejection fraction in obese patients upon admission to the hospital.
6. Characterize the severity and topical characteristics of congestion and compare with the phenotypes of acute decompensation of heart failure.
7. Assess adverse in-hospital outcomes and outcomes 6 months after hospital discharge and identify factors associated with them.
8. Conduct a clinical and instrumental examination of patients diagnosed with compensated and decompensated HFpEF, verified by echocardiography at rest, as well as in patients with HFpEF verified after an additional diastolic stress test with assessment of intracardiac hemodynamics.
9. Analyze the serum concentrations of biochemical markers associated with cellular stress (heat shock proteins) in these groups of patients, as well as in the control group of apparently healthy people.
10. Conduct an analysis of associations of biomarker levels with clinical characteristics of patients, the presence of comorbid diseases, including obesity, as well as with data from instrumental examination methods
11. Assess the diagnostic capabilities of HFpEF, defined by various criteria, based on the concentration of the new biomarkers studied

STUDY DESIGN:

Descriptive, open-label, observational study, randomization procedure not planned.

STAGES OF RESEARCH:

1. hospital: creating a patient database followed by:

It is planned to create a database, followed by:

* filling out the consent
* creation of a research registration card indicating:

  * Gender
  * Age;
  * Smoking;
  * Previous diagnosis of chronic heart failure;
  * Hyperthermia;
  * Time from the onset of symptoms to hospitalization, days;
  * Taking diuretics on an outpatient basis;
  * Taking renin-angiotensin aldosterone blockers on an outpatient basis;
  * Taking type 2 sodium glucose cotransporter inhibitors on an outpatient basis;
  * Taking anticoagulants on an outpatient basis;
  * Taking beta blockers on an outpatient basis;
  * Reception of mineralocorticoid receptor antagonists) on an outpatient basis;
  * Taking non-steroidal anti-inflammatory drugs on an outpatient basis,
  * Alcohol abuse,
  * Limited mobility
  * Arterial hypertension
  * Coronary heart disease,
  * Chronic obstructive pulmonary disease,
  * Body mass index,
  * Vaccination,
  * Valvular heart defects,
  * Diabetes;
  * Oncological diseases,
  * Chemotherapy,
  * Gastrointestinal pathology,
  * Chronic kidney disease)
  * Chest X-ray;
  * Natriuretic peptide on admission;
  * B-lines upon admission;
  * Therapy with intravenous diuretics;
  * Oral diuretic therapy;
  * Renin-angiotensin-aldosterone system blockers permanently;
  * Type 2 sodium glucose cotransporter inhibitors
  * Anticoagulant therapy in the hospital;
  * Height;
  * Weight;
  * Orthopnoea
  * Swelling of the neck veins;
  * Edema of the lower extremities;
  * Hepatomegaly;
  * Total water content;
  * Total fat content;
  * Left ventricular ejection fraction;
  * Pulmonary arterial systolic pressure,
  * Relative wall thickness;
  * Thickness of epicardial fat
  * Inferior vena cava, mm
  * Collapse of the Inferior vena cava
  * Diameter of the renal vein, mm
  * Portal vein diameter, mm
  * Enzyme immunoassay of heat shock proteins.
  * Analysis of routine biochemical parameters.
  * Duration of hospitalization, days.

Stage 2 - determining the nearest outcomes - In-hospital outcomes: death with indication of the cause of death, transfer with aggravation to another department of the hospital, discharged

Stage 3 - assessment of long-term outcomes after 6 months, which includes:

* creating a phone contact card
* determine vital status (alive/died) by telephone, and for the deceased, determine the cause of death and date, place of death, for the living - the number of hospitalizations over the past 6 months.
* identify repeated hospitalizations over the past period.
* entering the received data into the created electronic database in the data register and conducting statistical analysis

EXPECTED RESULTS The results obtained will allow us to evaluate the characteristics of the course and outcomes of the disease in Moscow patients, depending on the phenotype of acute decompensation of HFpEF, hospitalized in the hospital during the study period. When studying a cohort of patients hospitalized for emergency reasons, it is expected to identify phenotypes of acute decompensation of HFpEF that affect the duration of hospitalization and the development of adverse outcomes in the hospital and long-term period of the disease.

The prospects for further use in clinical practice of analysis of circulating levels of heat shock proteins in combination with other clinical and instrumental methods will be analyzed. Based on the data obtained, it is planned to develop laboratory and instrumental algorithms for additional assessment in patients with HFpEF.

ELIGIBILITY:
Inclusion Criteria:

All patients hospitalized with a clinical picture of acute decompensation of heart failure (shortness of breath, orthopnea, clinical signs of "cardiac asthma" and/or "pulmonary edema") in the city clinical hospital named after. V.V. Veresaeva, Moscow. Patients with a confirmed diagnosis in accordance with instrumental (EchoCG) and/or laboratory criteria.

Exclusion Criteria:

Refusal to sign informed consent to participate in a clinical trial and to process personal data.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Generic Moscow population
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Amount of secondary hospitalisations | 6 months
  Hospitalisations with decompensation of HFpEF

SECONDARY OUTCOMES:
Amount of hospitalisations with acute coronary syndrome | 6 months
Amount of hospitalisations with stroke | 6 months
Amount of hospitalisations with pulmonary embolism | 6 months
Amount of other cardiovascular events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yury Timfeev, PhD, Principal Investigator — National Medical Research Center for Therapy and Preventive Medicine; Olga Dzhioeva, MD, Study Director — National Medical Research Center for Therapy and Preventive Medicine; Timofei Vedenikin, Principal Investigator — Moscow State Clinical Hospital named after V.V. Veresaev
Locations (2):
- Russia (2):
  - Moscow State Clinical Hospital named after V.V. Veresaev, Moscow
  - National Medical Research Center for Therapy and Preventive Medicine, Moscow

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Timofeev YS, Kiselev AR, Dzhioeva ON, Drapkina OM. Heat Shock Proteins (HSPs) and Cardiovascular Complications of Obesity: Searching for Potential Biomarkers. Curr Issues Mol Biol. 2023 Nov 23;45(12):9378-9389. doi: 10.3390/cimb45120588. PMID 38132434
- [Result] Rogozhkina E.A., Vedenikin T.Yu., Timofeev Yu.S., Ivanova A.A., Afaunova A.R., Dzhioeva O.N., Drapkina O.M. Comparative assessment of venous congestion severity and hospitalization outcomes in patients with acute decompensated heart failure with preserved ejection fraction. Russian Journal of Cardiology. 2024;29(7):5977. (In Russ.) https://doi.org/10.15829/1560-4071-2024-5977. EDN: RGBFNE
- [Result] Timofeev Yu.S., Afaunova A.R., Ivanova A.A., Vedenikin T.Yu., Dzhioeva O.N., Metelskaya V.A., Pokrovskaya M.S., Drapkina O.M. Interaction of serum heat shock proteins' levels with the severity of venous congestion in patients with acute decompensated heart failure with preserved ejection fraction. Cardiovascular Therapy and Prevention. 2024;23(6):4037. (In Russ.) https://doi.org/10.15829/1728-8800-2024-4037. EDN: HXKJTD
- [Result] Timofeev Yu.S., Vedenikin T.Yu., Afaunova A.R., Zamyatin R.A., Metelskaya V.A., Dzhioeva O.N., Ivanova A.A., Neshkova E.A., Pokrovskaya M.S., Drapkina O.M. Heat shock proteins in the assessment of the course and prognosis of heart failure with preserved ejection fraction. Russian Journal of Cardiology. 2025;30(4):6317. (In Russ.) https://doi.org/10.15829/1560-4071-2025-6317. EDN: YHFXWZ
- [Result] Timofeev Yu.S., Metelskaya V.A., Ivanova A.A., Dubovskaya N.I., Rogozhkina E.A., Vedenikin T.Yu., Zamyatin R.A., Borisova A.L., Dzhioeva O.N., Drapkina O.M. Serum biochemical profile in patients with decompensated heart failure with preserved ejection fraction depending on obesity. Cardiovascular Therapy and Prevention. 2025;24(7):4453. (In Russ.) https://doi.org/10.15829/1728-8800-2025-4453. EDN: TEWGYU